CLINICAL TRIAL: NCT06769542
Title: The Effect of Micro Teaching Method on Nursing Students' Psychomotor Skills, Attitudes, Self-Efficacy and Clinical Stress Level: Randomized Controlled Trial
Brief Title: The Effect of Micro Teaching Method on Nursing Students' Psychomotor Skills, Attitudes, Self-Efficacy and Clinical Stress Level
Acronym: Microteach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Feride Kaplan
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Nursing Students
Keywords: Microteaching,; Clinical stress,; Psychomotor skills,; Self-efficacy,; Nursing Students

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Micro Teaching method
  Interventions: Behavioral: Experimental (micro teaching)
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Experimental (micro teaching) — The experimental group was taught using the micro-teaching method for 8 weeks. Psychomotor skills for drug administration were performed on models. Video recordings were taken while the students were performing the skills. These videos were evaluated by the instructor and the students and the students were given the opportunity to see their own mistakes. During 8 weeks, each student was given the opportunity to perform the applications and evaluate themselves. In addition, activities for drug applications were carried out with students within the scope of small group work. Micro teaching with 4 groups of 8 students was applied for 8 weeks.
  Arms: Experimental Group

SUMMARY:
Objective: This study was conducted to evaluate the effect of the micro-teaching method on nursing students' psychomotor drug administration skills, attitudes towards clinical practice, self-efficacy and clinical stress levels.

Method: The study was conducted as a pretest-posttest randomised controlled experimental research model. It was conducted between September 2023 and December 2024 at Kahramanmaraş Sütçü İmam University, Afşin School of Health, Department of Nursing. The population of the study consisted of all first year students of the Nursing Department. The sample consisted of 64 students (experimental group = 32, control group = 32) determined by power analysis. The following instruments were used to collect the data: "Drug administration skills assessment lists", "Attitudes towards clinical practice in nursing students scale", "Academic self-efficacy scale" and "Clinical stressor perception scale". During the first 3 weeks of the study, the topics related to drug administration were explained to the experimental and control groups 2 days a week for 6 hours each, and the applications were demonstrated using the demonstration method. From the 4th week of the study, the experimental group was taught using the micro-teaching method for 8 weeks.

DETAILED DESCRIPTION:
Micro-teaching method is a very valuable teaching method in psychomotor skills training in terms of providing feedback to the student, giving the opportunity to realise and correct their mistakes in line with this feedback, providing the opportunity to evaluate themselves while practising, creating a laboratory environment, eliminating the complexity of the application, ensuring active participation in the lesson, reducing anxiety, increasing self-confidence, gaining more experience by controlling the applications, and enabling even difficult applications to be performed.

In addition to the advantages of the micro-teaching method in itself, the fact that it is cost-effective, that students make active teaching in small groups, that lesson plans are made again until the applications are learnt, that peers and the instructor provide feedback during these applications, and that students have the opportunity to make their own self-evaluations with the videos recorded for skill applications suggest that it is an effective method in nursing skills training.

ELIGIBILITY:
Inclusion Criteria:

* To take the Nursing Principles course for the first time,
* To approve the evaluation and video recording of their practices,
* Volunteering to participate in the research,
* Being over 18 years old.

Exclusion Criteria:

* To have received an education related to parenteral applications other than basic nursing education,
* Not wanting/not being able to use micro-teaching method
* Absenteeism in the theoretical course,
* Wanting to leave during the research process,
* Not graduating from vocational high schools related to health departments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Effect of micro teaching on psychomotor skill level | 2 month
  In order to evaluate the psychomotor skill level of the students in the groups, drug administration skills of each student were evaluated individually by the researcher and independent observer and skill checklists for drug administration were filled.
  After the 8-week teaching plan with the micro-teaching method, the psychomotor skill levels of the students were evaluated by filling out the skill checklists for drug applications.
Effect of micro teaching on attitude for clinical practices | 2 month
  In order to evaluate the attitude for clinical practices in nursing students used the 'Attitude Scale for Clinical Practices in Nursing Students'. A score between 26 and 130 can be obtained from the scale, the higher the score, the more favourable the attitude.Students were asked to fill in the scale for pre-test and post-test measurement.
Effect of micro teaching on attitude for academic self efficacy | 2 month
  In order to evaluate the attitude for academic self efficacy in nursing students used the 'Academic Self-Efficacy Scale for Nursing Students'. In the 14-item, five-point Likert-type scale, a score ranging from 1 to 5 is obtained for the answer to each question and all of them consist of positive items. The increase in the score indicates an increase in academic self-efficacy. Students were asked to fill in the scale for pre-test and post-test measurement.
Effect of micro teaching on attitude for clinical stressor perceptions | 2 month
  In order to evaluate the clinical stressor perceptions in nursing students used the 'Scale of Clinical Stressor Perceptions of Nursing Students'. The scale consists of 22 items and 6 sub-dimensions (inappropriate situations in the clinical environment, inappropriate behaviours of the instructor, academic performance of the instructor, attitude of the instructor towards education, insufficient knowledge and skills of the student, concerns about nursing care). A score between 22 and 110 points can be obtained from the scale. A decrease in the score indicates a decrease in stressor perceptions.
  Students were asked to fill in the scale for pre-test and post-test measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Hakime Aslan, Principal Investigator — Inonu University
Locations (1):
- Hakime Aslan, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aslan H, Celik H, Kaplan F. The Relationship Between Palliative Care Nurses' Frequency of Providing Spiritual Care and Their Job Satisfaction: A Cross-Sectional Study. J Palliat Care. 2025 Jul;40(3):195-204. doi: 10.1177/08258597241301988. Epub 2024 Dec 18. PMID 39692344